CLINICAL TRIAL: NCT05632016
Title: The Impact of Erector Spinae Block (ESP)on Neurophysiological Monitoring in Patients Undergoing Scoliosis Repair Under TIVA
Brief Title: The Impact of ESP on Neurophysiological Monitoring in Scoliotic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU R193/2022
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Neurophysiological Monitoring Under TIVA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group N (No Intervention): patients will not receive erector spinae block (ESP)
- group E (Active Comparator): patients will receive bilateral bilevel erector spinae block (ESP)
  Interventions: Procedure: erector spinae block (ESP)

INTERVENTIONS:
Procedure: erector spinae block (ESP) — the erector spinae plane block will be performed bilaterally using a high-frequency-curved ultrasound transducer (Mindray 35C50EB, China) placed in a longitudinal orientation 3 cm lateral to the spinous process at two different levels, one above the angle of kyphosis at T8- T10 and another below the angle of kyphosis at L3. An 8- cm 22-gauge block needle (EchoStim; Benlan Inc, Oakville, Canada) is inserted in a cephalad-to-caudad direction until the tip lay in the interfascial plane below erector spinae muscle, the block will be performed by injection of 10 mL of bupivacaine at each point.A total volume of 40 ml of diluted bupivacaine with a total dose of 3mg/kg with variable concentrations according to body weight will be given for each patient.
  Arms: group E

SUMMARY:
Scoliosis surgery requires intraoperative neuromonitoring. Electrophysiological monitors used include somatosensory evoked potentials (SEPS) and motor-evoked potentials (MEPS). MEPS are a measured muscular contraction produced by stimulation of the motor cortex via electrodes to the scalp. Evoked electromyography (EMG) of pedicle screws allows for evaluation of potential injury from incorrect screw placement. Anaesthetic agents: Volatile agents produce dose-related decreases in amplitude of MEPs. MEPs are also stopped with the use of neuromuscular blockade (NMB). It is accepted that an initial dose of a NMB agent will be metabolised before monitoring is required. Therefore a TIVA technique is the recommended anaesthetic technique for this procedure. Propofol has been shown to attenuate MEP signals and should be kept in mind. This effect can be mitigated with the use of Ketamine which increases SEP and MEP amplitudes. Benzodiazepines as well as opioids (including intrathecal opioids) have been shown to have minimal effect on signals. α2 agonists attenuate MEP amplitudes (3).

Accordingly, the goals of spine correction surgery include hemodynamic stability with no interference in neuromonitoring and optimal pain control. Multimodal analgesia is recommended in the preoperative intraoperative and postoperative periods. Intrathecal morphine has been shown to reduce pain scores and allow for improved postoperative analgesia. Remifentanil infusions are used to reduce propofol requirements thus improving neuromonitoring. Hyperalgesia has been noted but various strategies can be used to mitigate this. Intravenous lignocaine and ketamine have been shown to reduce opioid requirements. The use of α2 agonists help to reduce opioid requirements but can attenuate neuromonitoring signals.

Postoperative administration of extensive amounts of opioids can cause well known side-effects, such as respiratory depression, sedation, pruritis, nausea, vomiting, and constipation. Ileus is also a common complication due to the nature of the surgery and opioid use in the perioperative period. Even with opioids, pain is not always sufficiently managed. Inadequate pain control increases cardiac and respiratory complications, delays mobilization, increases the length of hospital stay and may increase the risk of developing a chronic pain syndrome . The above mentioned complications indicate the need for a novel regional anesthesia techniques. Until recently, regional anesthesia techniques have not been used on a regular basis in spine surgery as an immediate postoperative neurological examination is required. This examination of the motor and sensory function of the spinal cord eliminates spinal and epidural analgesia as suitable pain treatments. Novel interfascial plane blocks, such as the erector spinae plane (ESP) block, generate regional analgesia without interference of spinal cord function and are therefore suitable for spinal surgery pain management .

An ESP block has a very low risk of complications, as sonoanatomy is easily recognizable and there are no structures in close proximity at risk of needle injury. The transverse process acts as an anatomical barrier and avoids needle insertion into the pleura or vessels, thus preventing a pneumothorax or hematoma. Moreover, the needle is relatively far from the vertebral canal, which means the risk of spinal cord injury is very low. It is applied preoperatively before skin incision as a preemptive analgesia so it suppresses chronic sensitization process. In addition, it may abolish the neuroendocrine stress response by decreasing release of the counterregulatory hormones like catecholamines the mechanism by which it may augment controlled hypotensive anaesthesia

ELIGIBILITY:
Inclusion Criteria:

* patients with American Association of Anesthesiologists up to III physical status undergoing scoliosis repair under TIVA.

Exclusion Criteria:

* Patients with an ASA status above III.
* patient or guardian refusal to participate, patients with multiple congenital anomalies.
* hypersensitivity or contraindication to the study drugs.
* severe restrictive pulmonary disease indicating postoperative ventilation.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The effect of ESP on neurophysiological monitoring | the whole intraoperative time
  the effect of ESP on SSEPs and MEPs during scoliosis repair

SECONDARY OUTCOMES:
Intra and postoperative analgesic effect of ESP | 24 hours
  total dose of intraoperative and postoperative analgesics

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt